CLINICAL TRIAL: NCT05446116
Title: Transfemoral Versus Transradial Partial Splenic Artery Embolization in Patients With Hypersplenism, a Randomized Controlled Trial
Brief Title: Transfemoral Versus Transradial Partial Splenic Artery Embolization in Patients With Hypersplenism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed M.A. Zaitoun, Associate Professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zu-IRB#9027/13-6-2021
Record Dates: First submitted 2021-10-19; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Hypersplenism
MeSH Terms: conditions — Hypersplenism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- femoral puncture (Active Comparator): Under local anaesthesia, the femoral artery was punctured and 6F sheath was inserted. Splenic artery was catheterized using 4- or 5-F catheters (Cobra C2 cat or Simmons II catheter Imager-Boston Scientific Natick, Massachusetts). Embolization was done using Embospheres (Biosphere Medical, Rockland, MA) 700-900 μ in diameter.
  Interventions: Procedure: partial splenic artery embolization
- Radial puncture (Active Comparator): The left radial artery was preferred due to shorter distance from the left wrist to the splenic artery in comparison to the right wrist; also the left radial access theoretically decreases the risk of cerebral emboli. Under local anaesthesia and ultrasound guidance, the radial artery was punctured and 5- or 6-F sheath was introduced. After sheath insertion, the radial cocktail (2.5 mg of verapamil, 100 μg of nitroglycerin, and 5,000 units of heparin) was injected through the sheath over one minute after dilution with 20 ml of blood to decrease the discomfort during injection.
  Interventions: Procedure: partial splenic artery embolization

INTERVENTIONS:
Procedure: partial splenic artery embolization — embolization of the splenic artery for the treatment of hypersplenism

SUMMARY:
The present study aimes at comparing the transradial and transfemoral approaches for partial splenic embolization in patients with hypersplenism.

DETAILED DESCRIPTION:
Since its development in 1979, partial splenic embolization (PSE) has been universally accepted to treat patients with hypersplenism in preference to surgical splenectomy. The spleen is the primary source of antibodies, lymphocyte production, and responsible for phagocytosis of white cells. Additionally, it plays an essential role in the immune system. Unlike splenectomy, partial splenic embolization (PSE) maintained partial splenic function and was thought to be an effective alternative to treat thrombocytopenia and leukopenia resulted from hypersplenism with fewer complications.

PSE is usually performed using a femoral artery approach that requires bed rest for a few hours. Recently, the transradial approach, with less obvious need for bed rest, has been more widely applied for cardiovascular intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hypersplenism and severe thrombocytopenia (platelet count < 50,000/mm3).
2. the functional status of the liver should be Child A or early B according to Child-Pugh classification (5-7 points) (albumin ≥ 2.8 g/dL, bilirubin ≤ 3 mg/dL, prothrombin time ≤ 4 or INR < 1.7, no ascites, no encephalopathy).
3. Eligible for both femoral and radial puncture.

Exclusion Criteria:

1. Patients referred for embolization as treatment of traumatic splenic injury.
2. Patients lost during follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Technical Success of the Procedure | Immediately after the procedure is complete
  The achievement of a single puncture allowing access to splenic artery without periprocedural complications.
Average number of punctures | Immediately after the procedure is complete
  Number of arterial punctures required to complete the procedure
Procedural time | Immediately after the procedure is complete
  The time interval from starting the anaethesia till completion of the procedure
X-ray exposure duration | Immediately after the procedure is complete
  Duration of flouroscopy exposure during the procedure
Length of hospital stay | 7 days
  Number of days that the patient will spend in the hospital after the procedure.
Complications at access site | 30 days
  Access site adverse events such as vessel thrombosis, pseudoaneurysm or bleeding.

SECONDARY OUTCOMES:
Procedural complications | 30 days
  Adverse events related to the procedure itself like splenic abscess, ascitis or portal vein thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed MA Zaitoun, MD, Principal Investigator — Zagazig University Radiology Department
Locations (1):
- Faculty of medicine, Zagazig university, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No